CLINICAL TRIAL: NCT06980116
Title: A Phase 1 Open-label, Multicenter, Dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of EXS73565 in Participants With Relapsed or Refractory B-cell Malignancies
Brief Title: Dose Determining Study of EXS73565 in Participants With Relapsed or Refractory B-Cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Exscientia AI Ltd., a wholly owned subsidiary of Recursion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Exscientia AI Limited (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXS73565-001; 2024-516869-36-00 (EU CTIS Number); 2022-003475-42 (EudraCT Number)
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Relapsed or Refractory B-cell Malignancies
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EXS73565 (Experimental)
  Interventions: Drug: EXS73565

INTERVENTIONS:
Drug: EXS73565 — EXS73565 oral administration

SUMMARY:
The purpose of this study is to characterize the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary antitumor activity of EXS73565 administered orally as a single agent in participants with relapsed/refractory B-cell malignancies.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥18 years at the time of signing the informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Histologically confirmed diagnosis of one of the following B-cell malignancies: chronic lymphocytic leukemia (CLL), including Richter's transformation from CLL, mantle-cell lymphoma, diffuse large B-cell lymphoma, follicular lymphoma, or marginal zone lymphoma.
* Participants that have relapsed after standard of care or have progressed during standard of care or are not suitable for standard of care therapy

Key Exclusion Criteria:

* Any medical or psychiatric condition that, in the view of the Principal Investigator, could jeopardize or would compromise the participant's safety or ability to participate in the study.
* Known central nervous system (CNS) malignancy or primary CNS lymphoma.
* Concurrent active or previous malignancy (other than the primary lymphoma/CLL for which the participant will be treated on this protocol within 5 years prior to randomization; participants with prior cancers may be enrolled with documented Sponsor approval.
* Received anticancer therapy, including chemotherapy, immunotherapy, radiation therapy (with the exception of palliative radiotherapy), biologic therapy, cancer-related hormonal therapy, or any investigational therapy within 21 days or 5 half-lives (whichever is longer) before the first dose of the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to 282 days
Dose-limiting toxicities (DLTs) of EXS73565-001 | Up to 21 days

SECONDARY OUTCOMES:
Time to Maximum Concentration (Tmax) of EXS73565-001 | Up to 253 days
Area Under the Concentration-time Curve from Time Zero to the Time of the Last Quantifiable Concentration AUC(0-last) of EXS73565-001 | Up to 253 days
Maximum Concentration (Cmax) of EXS73565-001 | Up to 253 days
Overall Response Rate (ORR) | Up to 434 days
Disease Control Rate | Up to 434 days
Progression Free Survival | Up to 434 days
Duration of Response | Up to 434 days
Time to Respond | Up to 434 days
Time to Progression | Up to 434 days

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (2):
  - Hospital Fundación Jiménez Diaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
- United Kingdom (2):
  - St James's University Hospital, Leeds
  - University Hospitals Plymouth NHS Trust, Plymouth

IPD SHARING:
Plan to Share IPD: No